CLINICAL TRIAL: NCT03506984
Title: High Intensity Interval Training Versus Inspiratory Muscle Training on Modulating Blood Rheology in Coronary Artery Disease Risk Factors
Brief Title: HIIT Versus IMT on Modulating Blood Rheology in CAD Risk Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Elbanna, lecturer assistance at faculty of physical therapy at Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Rana Elbanna
Record Dates: First submitted 2018-03-15; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease, Early-Onset
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Participants will randomely divided into two equal groups. Group (A) will receive a programe of high intensity interval training 30-40 minutes three times per week for one month.the participant will start cycling slowly for five minute without resistance at the beginning of the exercise as warming up, then the active phase will last 20-30 minutes, then decrease the speed with no resistance at the end of the exercise as cooling down. The participant will be closely monitored by the handheld telemetry. Group (B) will receive a program of inspiratory muscle training by using the threshold based inspiratory muscle trainer for 10-15 minutesonce daily with frequency three times per week for four weeks.
Who Masked: Participant
Masking Description: the participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): the participant will do a program of inspiratory muscle training for 10-15 minutes once daily using Threshold Inspiration Muscle Training Device
  Interventions: Device: Threshold Inspiration Muscle Training Device
- Group B (Experimental): the participant will start cycling slowly for five minutes without resistance at the beginning of the exercise as warming up, then the active phase will last 20-30 minutes, then decrease the speed with no resistance at the end of the exercise as cooling down using Electronic Bicycle Ergometer
  Interventions: Device: Electronic Bicycle Ergometer

INTERVENTIONS:
Device: Threshold Inspiration Muscle Training Device — Threshold based trainer is a small handled device.It includes a mouthpiece and a calibrated spring loaded valve. The valve control a constant inspiratory pressure training load and the patient must generate a suffient inspiratory pressure in order for the inspiratory valve to be opened and allow the air to be inhaled. The amount of resistance can be adjusted by varying the compression of the spring-loaded valve. Adjustment from 9cmH2o to 41cmH2o.
  Other Names: respironics,cedarGrove,NJ 07009-1201 Made in U.S.A
  Arms: Group A
Device: Electronic Bicycle Ergometer — Electronic Bicycle equipped with electronic break, display screen, adjustable seat, handle bar and foot straps will be used in High interval intensity training.
  Other Names: Biodex LBC, made in New York
  Arms: Group B

SUMMARY:
Participants had randomly divided into two equal groups. Group (A) had received a program of high intensity interval training 30-40 minutes three times per week for one month. The participant will start cycling slowly for five minute without resistance at the beginning of the exercise as warming up, then the active phase will last 20-30 minutes, then decrease the speed with no resistance at the end of the exercise as cooling down. Group (B) will receive a program of inspiratory muscle training by using the threshold based inspiratory muscle trainer for 10-15 minute daily with frequency three times per week for four weeks.

DETAILED DESCRIPTION:
Training Procedure for group (A):

1. Each participant had signed a consent form after receiving a detailed explanation about the procedure.
2. BMI had been measured body weight(Kg) and height (m2)

   a. BMI= body weight (Kg)/ height (m2).
3. Resting pulse rate had been measured to the participant three successive times then the mean had to be taken.
4. A blood sample had been taken by a nurse in a heparinized tube and delivered to lab within six hours.
5. The participant had been asked to walk as quickly as he could in a 30-meter pre-measured flat walking area with interval markings every three meters for six minutes. Cones or brightly colored tape to mark boundaries of the walkway with cones placed at the beginning and end of the 30-meter boundary to indicate turns. (Actual distance). (BALKE 1963)
6. Teaching the participant had been reached how to perform high interval training exercise.
7. The load had been determined according to maximum heart rate obtained from cardiopulmonary exercise testing performed by cardiologist.
8. high intensity (85% - 95% MHR) and the interval period (60% - 75% MHR) .(Gibala et al. 2006)
9. The participant's started by five minutes warming up on the bicycle ergometer with no resistance as shown in fig (8).
10. Then one minute of high intensity training followed by one and half minute of low intensity training for 20 to 30 minutes.
11. Finally, a five minutes of cooling down with no resistance had performed.
12. Post treatment evaluation had been done using step three, four and step five.

Training Procedure for group (B):

1. Each participant had signed a consent form after receiving a detailed explanation about the procedure.
2. BMI had been measured body weight(Kg) and height (m2)

   a. BMI= body weight (Kg)/ height (m2).
3. Resting pulse rate had been measured to the participant three successive times then the mean had to be taken.
4. A blood sample had been taken by a nurse in a heparinized tube and delivered to lab within six hours.
5. The participant had been asked to walk as quickly as he could in a 30-meter pre-measured flat walking area with interval markings every three meters for six minutes. Cones or brightly colored tape to mark boundaries of the walkway with cones placed at the beginning and end of the 30-meter boundary to indicate turns. (Actual distance). (BALKE 1963)
6. Teaching the participant had been teached how to use the threshold based Inspiratory muscle trainer device.
7. The load had been determined according to 10 maximum repetitions (10RMax).
8. The intensity had been 60% to 80% of the participant's maximal effort.(Enright & Unnithan 2011)
9. The Inspiratory Muscle Trainer had been applied for (10 to 15) minutes once daily with frequency three times per week for four weeks as shown in fig (9).
10. Post treatment evaluation had been done using step three, four and step five.

ELIGIBILITY:
Inclusion Criteria:

1. They will be 45-55 years old participants of males.
2. All of them had body mass index more than 30 kg/m2.
3. All of them were diagnosed as diabetic persons for at least 5 years.
4. All of them were diagnosed as a mild to moderate hypertensive persons for at least 5 years.
5. All of them had a reduction in walking capacity in relation to their height, age and body mass index (BMI).

Exclusion Criteria:

1. Unstable cardiac condition.
2. Patient who were on beta blocker.
3. Uncontrolled diabetes mellitus.
4. Mentally unstable person.
5. Patient with intermittent claudication.

Ages: 45 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-25 (Estimated); Study Completion 2018-05-03 (Estimated)

PRIMARY OUTCOMES:
Compare between the effect of High Intensity Interval Training versus Inspiratory Muscle Training on modulating lipid profile ( cholesterol level mg/dl, triglyceride mg/dl, LDL mg/dl and HDL mg/dl) by using the blood analyzer in CAD risk factors | after 4 weeks of the trial application
  Comparison between the effect of High Intensity Interval Training versus Inspiratory Muscle Training on modulating lipid profile which composed of ( cholesterol level mg/dl, triglyceride mg/dl, LDL mg/dl and HDL mg/dl) by using the blood analyzer (Photometer, 5010, boehinger) in Coronary Artery Disease risk factors

SECONDARY OUTCOMES:
Effect of high intensity interval training and Inspiratory Muscle Training on 6 minutes walking test by meter | after 4 weeks of the trial application
  Effect of high intensity interval training and Inspiratory Muscle Training on 6 minutes walking test by meter
Compare between the effect of High Intensity Interval Training versus Inspiratory Muscle Training on modulating hematocrit value by using the blood analyzer in CAD risk factors | after 4 weeks of the trial application
  Comparison between the effect of High Intensity Interval Training versus Inspiratory Muscle Training on modulating hematocrit value (The proportion of the blood that consists of packed red blood cells) % by using the blood analyzer (Photometer, 5010, boehinger) in Coronary Artery Disease risk factors
Effect of high intensity interval training and Inspiratory Muscle Training on pulse rate (beat/min) | after 4 weeks of the trial application
  Effect of high intensity interval training and Inspiratory Muscle Training on pulse rate (beat/min)
Effect of high intensity interval training and Inspiratory Muscle Training on modified BORG scale by meter | after 4 weeks of the trial application
  Effect of high intensity interval training and Inspiratory Muscle Training on modified BORG scale by meter

CONTACTS AND LOCATIONS:
Overall Officials: Rana H Elbanna, master, Principal Investigator — lecturer assistance at faculty of physical therapy at Cairo University
Locations (1):
- Ibri hospital, Ibri, Al Dhahra, Oman

IPD SHARING:
Plan to Share IPD: Undecided
not decided